CLINICAL TRIAL: NCT05440669
Title: The Effect of White Noise on Pain and Stress Level in Nasal Cpap Application
Brief Title: White Noise in Nasal Cpap Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ARZU SARIALİOĞLU, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/448
Record Dates: First submitted 2022-06-22; First posted 2022-07-01 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Nasal Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- White Noise (Experimental): white noise will reduce pain and stress
  Interventions: Behavioral: white noise
- control (No Intervention): white noise will not reduce pain and stress

INTERVENTIONS:
Behavioral: white noise — white noise will reduce pain and stress in nasal cpap application
  Arms: White Noise

SUMMARY:
The aim of this study is to determine the effect of white noise application on the pain and stress level of newborns receiving oxygen support via nasal CPAP in the Neonatal Intensive Care Unit. The research is a randomized controlled trial. The population of the study will be infants aged 0-28 days who were hospitalized for treatment in Şanlıurfa Training and Research Hospital between July and December 2022. The research sample; Babies of families who are hospitalized in the Neonatal Intensive Care Unit on the specified dates and meet the research criteria and volunteer to participate in the research will be formed. "Survey Form", "Follow-up Form" and "ALPS Neo Neonatal Pain and Stress Assessment Scale", White Noise, MP 3 Player, and Sound Decibel Measuring Device will be used to collect data.

DETAILED DESCRIPTION:
Type of Study: The study is planned experimentally with a randomized control group.

Place and Time of the Research: The research will be carried out between June-December 2022 in Şanlıurfa Training and Research Hospital Neonatal Intensive Care Unit. There are 130 incubators in total, with 53 beds at the 2nd level and 54 beds at the 3rd level. 55 respirators, 4 fully equipped transport incubators with respirators, isolation room, 4 hypothermia devices, 2 Aeeg devices etc. are available. Treatments that can be performed in the Neonatal Intensive Care Unit; respiratory support (ventilator therapy), thoracic tube insertion, blood exchange, total parenteral nutrition, phototherapy, percutaneous catheter applications, patient transport with 24-hour incubators with breathing apparatus, dialysis catheter insertion and follow-up, colostomy care, etc. are treatments. A total of 133 nurses work.

Population and Sampling of the Study: The population of the study will consist of infants aged 0-28 days who will receive oxygen therapy in nasal CPAP by being hospitalized in the Newborn Intensive Care Unit of Şanlıurfa Training and Research Hospital between July and December 2022 due to respiratory distress.

In this study, "prior power analysis" was used to determine sample adequacy. In the power analysis used, "Cohen's standard effect size reference technique" was chosen. In this case, for the t-test in independent groups, it was determined that if the study was advanced with 80 participants in two groups with 40 participants in each group, 80% power could be reached at a significance level of 0.05, at a 95% confidence interval. Against the possibility of data loss, it was decided to collect data from a total of 100 individuals by adding 10% more backup sample to this number. In order to ensure randomization, babies who meet the criteria will be taken to the control group, who are in the first week, and to the experimental group, respectively, and this cycle will be continued until the end of the research, and randomization will be ensured.

Inclusion Criteria for Research

* 38-40 weeks of gestation
* Receiving oxygen support in nasal CPAP
* Not taking opioids or sedatives 4 hours before the procedure.

Data Collection Tools to be Used in the Study: : "Survey Form, Neonatal Pain and Stress Assessment Scale, Follow-up Form, White Noise, MP 3 Player, and Sound Decibel Measuring Device" will be used to collect research data.

Questionnaire Form: In this form, which was prepared by the researcher by examining the literature; There will be questions about the introductory features of the newborn.

ALPS Neo Neonatal Pain and Stress Rating Scale: The "ALPS Neo Neonatal Pain and Stress Rating Scale" was developed in 2014, based on the individualized developmental care of the newborn, in order to evaluate pain and stress in premature and term newborns. In 2017, this scale was adapted to Turkish and its validity and reliability study was conducted. The scale is a 3-point Likert-type scale consisting of 5 parameters: "newborn's facial expression, breathing pattern, tone of the extremities, hand/foot activities, and activity level". As the scores increase, pain and stress increase in the newborn. As a result of the evaluation, "3-5 points indicate the presence of mild pain and stress, and more than 5 points indicate the presence of severe pain and stress".

Follow-up Form: It is a form used to record the newborn's cardiorespiratory parameters (peak heart rate, oxygen saturation), ALPS Neo pain scale, and crying time evaluated during nasal CPAPP.

Intervention Tool to be Used in Research White noise: Dr. Orhan Osman to calm the babies. It was prepared by making use of the album "Happy Baby" prepared by Harvery KARP, which consists of only intrauterine sounds.

Sound decibel meter: It will be used to determine the sound level of the white noise concert. The application will be made so that the level in the environment is 45-55 dB.

Mp3 player: It will be used for listening to white noise. Data Collection The research data will be collected from the babies of the families who agreed to participate in the research after the researcher gave the parents of the patients preliminary information about the research (the purpose of the research, why the research was conducted, the attempt to relieve the neonatal pain with a non-pharmacological method, etc.) and after their written consent was obtained. The purpose of making the patient listen to white noise; It is to reduce the pain and stress level of the procedure to a minimum level by ensuring that the patient calms down.

Experimental Group: Babies in this group will be listened to white noise for five minutes before nasal CPAP is applied.5. After 1 minute, nasal CPAP application will be started. White noise will continue to be listened during the application. Before the application, during the application, after the patient will be evaluated with the ALPS-Neo Neonatal Pain and Stress Rating Scale and the scale and follow-up form will be filled.

Control Group: Nasal CPAP will be routinely applied to babies in this group and the patient will be evaluated with the ALPS Neo Neonatal Pain and Stress Rating Scale before, during and after the procedure, and the scale and follow-up form will be filled.

Evaluation of Data Evaluation of statistics will be done by blinding method. Data will be collected by the researcher. The analysis of the data will be done by the statistician. The data will be sent after making sure that the data is coded in a way that preserves the blinding (without knowing which of the control and experimental groups). SPSS package program will be used for data analysis. The normality distribution of the data will be determined by the Kurtosis and Skewness coefficients. For the analysis of the data, "t-test for normally distributed measurements in the comparison of paired groups with numbers, percentages, mean and standard deviations, and Mann Whitney U test for non-normally distributed measurements" will be used. In the comparison of multiple groups, "Analysis of variance" will be used for normally distributed measurements, and Kruskall Wallis test for non-normally distributed measurements.

Ethical Principles of Research In order to carry out the research, official permission will be obtained from the relevant institution with ethical approval. The purpose of the study will be explained to the parents of the babies with the research group criteria, the questions asked will be answered and their verbal and written consent will be obtained. Parents will be informed that the data collected during the research will be processed anonymously, confidentially, and will not be used outside of the study in question, and that they can leave the study whenever they wish. Since the research is based on the use of data obtained from humans, and therefore, due to the necessity of observing personal rights, the relevant ethical principles "Informed Consent", "Volunteerism" and "Protection of Confidentiality" will be followed.

ELIGIBILITY:
Inclusion Criteria:

* 38-40 weeks of gestation
* Receiving oxygen support in nasal CPAP
* Not taking opioids or sedatives 4 hours before the procedure

Exclusion Criteria:

* Not at 38-40 weeks of gestation
* Not receiving oxygen support in nasal CPAP
* Taking opioids or sedatives 4 hours before the procedure

Ages: 38 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-06-19 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
ALPS Neo Neonatal Pain and Stress Rating Scale | 9 MONTHS
  The "ALPS Neo Neonatal Pain and Stress Rating Scale" was developed in 2014, based on the individualized developmental care of the newborn, in order to evaluate pain and stress in premature and term newborns. In 2017, this scale was adapted to Turkish and its validity and reliability study was conducted. The scale is a 3-point Likert-type scale consisting of 5 parameters: "newborn's facial expression, breathing pattern, tone of the extremities, hand/foot activities, and activity level". As the scores increase, pain and stress increase in the newborn. As a result of the evaluation, "3-5 points indicate the presence of mild pain and stress, and more than 5 points indicate the presence of severe pain and stress".

CONTACTS AND LOCATIONS:
Overall Officials: ARZU SARIALİOĞLU, PHD, Study Director — Ataturk University
Locations (1):
- Ataturk University Nursing of Faculty, Erzurum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE ARTICLE IS INTENDED TO BE SHARED AFTER IT IS PUBLISHED

REFERENCES:
- [Derived] Gokturk G, Sarialioglu A. Effect of white noise during nasal continuous positive airway pressure application on newborn's pain and stress levels, physiological parameters, and crying durations: A randomized controlled study. J Pediatr Nurs. 2024 Sep-Oct;78:e330-e337. doi: 10.1016/j.pedn.2024.07.022. Epub 2024 Jul 26. PMID 39060170